CLINICAL TRIAL: NCT02165150
Title: Development, Application , and Evaluation of the Senior Elastic Band (SEB) Exercise Program for Elderly Residents in Long-term Care Facilities
Brief Title: Senior Elastic Band (SEB) on Institutional Elders
Acronym: SEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Kuei-Min Chen, Ph.D., RN., Professor, Kaohsiung Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FYH-IRB-098-12-02; NSC99-2628-B-037-066-MY3 (Other Grant/Funding Number: National Science Council)
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Institutional Older Adults
Keywords: Elastic Band; Institutional Elders; Functional Fitness; Sleep Quality; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wheelchair-bound Senior Elastic Band (Experimental): WSEB interventions three times per week, 40 minutes per practice
  Interventions: Other: Wheelchair-bound Senior Elastic Band exercise program
- Control (No Intervention): routine care

INTERVENTIONS:
Other: Wheelchair-bound Senior Elastic Band exercise program — three times per week, 40 minutes per practice
  Arms: Wheelchair-bound Senior Elastic Band

SUMMARY:
The goals of this research project are: 1) to develop and evaluate the safety and feasibility of the Senior Elastic Band (SEB) exercise program for elderly residents in long term care facilities, 2) to evaluate the long-term effects of the SEB on physical functional fitness and sleep quality of elderly residents in long term care facilities, and 3) to investigate the compliance of elderly residents with long-term SEB exercises.

DETAILED DESCRIPTION:
A three-year, longitudinal, triangulation research method will be used. The study purpose of the first year is to develop a safe and appropriate SEB program for the elderly residents in long term care facilities using Delphi survey with a panel of 12 experts and pilot-testing on a group of 15-20 elderly residents in long term care facilities. In the second year of the study, a quasi-experimental, non-equivalent control group design will be used to evaluate the effects of the SEB exercise program on the physical functional fitness (cardiovascular-respiratory function, body flexibility, muscle power/muscle endurance, and balance) and sleep quality of elderly residents in long term care facilities. Through the convenience sampling strategy, a total of four long term care facilities with approximately 120 elders in Kaohsiung will be recruited and randomly assigned based on the resided facilities to a SEB experimental group or a waiting-list control group. The subjects in the experimental group will receive the SEB interventions lead by the certified instructors, three times per week, 40 minutes per practice for six months; the subjects in the waiting-list control group will remain regular daily activities in the facilities. All subjects will receive one pre-test and two post-tests three months apart during the study. In the third year, the elderly participants will continue practicing the SEB guided by a VCD for another nine months, and the compliance of the participants toward regular SEB exercise and its long-term effects on the physical functional fitness and sleep quality outcomes will be tested with additional three post-tests, three months apart.

ELIGIBILITY:
Inclusion Criteria:

* elderly residents aged 65 and over
* Mandarin or Taiwanese speakers
* have been living in the facility for at least 3 months
* able to stand alone without assistive devices
* cognitively alert and able to verbally state their name, address, and answer questions.

Exclusion Criteria:

* participants with severe and acute cardiovascular, musculoskeletal, or pulmonary illnesses

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in physical functional fitness at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  including cardiovascular-respiratory function, body flexibility, muscle power/muscle endurance, and balance

SECONDARY OUTCOMES:
Change from baseline in sleep quality at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  measured by PSQI
Change from baseline in depression at 3, 6, 9, 12, 15 months | participants will be followed for 15 months
  measured by Taiwanese Depression Questionnaire (TDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Kuei-Min Chen, Ph.D., Principal Investigator — Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan